CLINICAL TRIAL: NCT03808818
Title: Implementing a Virtual Tobacco Treatment in Community Oncology Practices: "Smoke Free Support Study 2.0"
Brief Title: Implementing a Virtual Tobacco Treatment for Cancer Patients in Community Oncology Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EAQ171CD; NCI-2018-02826 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ171CD (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EAQ171CD (Other: DCP); EAQ171CD (Other: CTEP); R01CA214427 (NIH)
Record Dates: First submitted 2019-01-08; First posted 2019-01-18 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma In Situ; Current Smoker; Malignant Neoplasm; Primary Neoplasm; Recurrent Neoplasm; Smoking Cessation
MeSH Terms: conditions — Carcinoma in Situ; Neoplasms; Recurrence; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (smoking assessment, quitting advice, Quitline referral) (Active Comparator): Patients receive an assessment of smoking status and provision of quitting advice through the screening and referral process, and are referred to the NCI Smoking Quitline.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Quality-of-Life Assessment
- Arm B (virtual counseling sessions, NRT) (Experimental): Patients receive an initial virtual counseling session with a study-designated tobacco treatment coach via MGH TeleHealth over 40 minutes and up to 10 more virtual counseling sessions over 15 minutes for approximately 6 months. Patients also receive up to 12 weeks of NRT (patch and lozenge combined or alone).
  Interventions: Drug: Nicotine Replacement; Other: Quality-of-Life Assessment; Other: Survey Administration; Other: Tobacco Cessation Counseling

INTERVENTIONS:
Other: Behavioral, Psychological or Informational Intervention — Receive information about tobacco cessation
  Arms: Arm A (smoking assessment, quitting advice, Quitline referral)
Drug: Nicotine Replacement — Given NRT patch or lozenge (or both)
  Other Names: Nicotine Replacement Therapy; NRT
  Arms: Arm B (virtual counseling sessions, NRT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies
  Arms: Arm B (virtual counseling sessions, NRT)
Other: Tobacco Cessation Counseling — Receive virtual tobacco cessation counseling
  Arms: Arm B (virtual counseling sessions, NRT)

SUMMARY:
This phase II trial studies how well smoking cessation treatment plans work in tobacco-dependent cancer patients when delivered virtually as part of their cancer care in community oncology practices. Virtual information and counseling sessions may help cancer patients quit smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the proportions of participants in the Enhanced Usual Care (EUC) and Virtual Tobacco Treatment (VIT) study arms with biochemically-verified 7-day point-prevalence abstinence from cigarettes at 6-months post enrollment.

SECONDARY OBJECTIVES:

I. Biochemically-verified 7-day point prevalence abstinence at 3-months follow-up.

II. Self-reported 7-day point prevalence cigarette abstinence at 3- and 6-months follow-up.

III. Significant reduction (> 50% reduction in reported number of cigarettes per day) in daily smoking from baseline to 3- and baseline to 6-months follow-up.

IV. Continuous (no self-reported smoking since last survey point) and sustained abstinence at 6 months (cotinine-verified at 3-months and 6-months).

EXPLORATORY OBJECTIVES:

I. To assess the potential effect of known and potential moderators on treatment effectiveness between the two arms.

II. To assess the processes of implementation and dissemination (acceptability, adoption, appropriateness, treatment fidelity, cost effectiveness, penetration/reach, and sustainability) of the investigator's intervention at community oncology sites.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A (Enhanced Usual Care [EUC]): Patients receive an assessment of smoking status and provision of quitting advice through the screening and referral process, and are referred to the National Cancer Institute (NCI) Smoking Quitline.

ARM B (Virtual Intervention Treatment [VIT]): Patients receive an initial virtual counseling session with a study-designated tobacco treatment coach via MGH TeleHealth over 40 minutes and up to 10 more virtual counseling sessions over 15 minutes for approximately 6 months. Patients also receive up to 12 weeks of nicotine replacement (NRT) (patch and lozenge combined or alone).

After completion of study, patients may be followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* STAFF ELIGIBILITY CRITERIA:
* Must be English speaking.
* Must be employed at NCI Community Oncology Research Program (NCORP) site for at least three months.
* PATIENT ELIGIBILITY CRITERIA STEP 0:
* Patient presenting with any type of cancer with a date of diagnosis within the past 4 months. Recurrence, diagnosed within the last 4 months, of tumors in patients with past cancer diagnoses will be considered eligible. Patients with a new primary cancer, diagnosed within the last 4 months, who have been treated previously for other types of cancer will also be considered eligible. ?In situ? cancers, diagnosed within the past 4 months, will also be considered eligible.
* Patient must be a current smoker. Current smoker is defined as any cigarette smoking (even a puff) in the past 30 days.
* Patient must be fluent in both, written and spoken, English or both, written and spoken, Spanish.
* Patient must have telephone, e-mail access, and have access to the internet with a camera-enabled device (e.g., smartphone, tablet, computer, laptop with a webcam/camera)

  * NOTE: The restriction to those with web and e-mail access is based on the primary intention of the study; to assess the implementation of the virtual intervention in the NCORP network.
* ELIGIBILITY CRITERIA STEP 1: Patient must still meet all criteria outlined in step 0.
* ELIGIBILITY STEP 2 (RANDOMIZATION): Patient must have completed baseline survey in Eastern Cooperative Oncology Group-American College of Radiology Imaging Network (ECOG-ACRIN) Cancer Research Group Systems for Easy Entry of Patient Reported Outcomes (EASEEPRO) within 1 month (30 days) of the date of informed consent (Step 1).

Exclusion Criteria:

* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 3 or above, or is deemed medically unable to participate by study investigators or oncology clinician (i.e., referral to hospice).
* Patient has no intention to receive their cancer care or monitoring at an NCORP community cancer site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse Park, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (42):
- United States (42):
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Carle on Vermilion, Danville, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Unity Hospital, Fridley, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Freeman Health System, Joplin, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - MultiCare Auburn Medical Center, Auburn, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Derived] Goshe BM, Rasmussen AW, Wagner LI, Sicks JD, Gareen IF, Carlos RC, Herman BA, Walter AW, Regan S, Levy DE, Mahon I, Muzikansky A, Neil JM, Lui M, Dilip D, Malloy L, Gonzalez I, Finkelstein-Fox L, McCann C, Perez E, Ostroff JS, Park ER. Study protocol for a hybrid type 1 effectiveness-implementation trial testing virtual tobacco treatment in oncology practices [Smokefree Support Study 2.0]. BMC Public Health. 2022 Jul 15;22(1):1359. doi: 10.1186/s12889-022-13631-w. PMID 35841024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients recruited between April 2019 and December 2022
Groups:
- EUC (Smoking Assessment, Quitting Advice, Quitline Referral): Enhanced usual care (EUC) participants receive an assessment of smoking status and provision of quitting advice through the screening and referral process, and are referred to the NCI Smoking Quitline.
  Behavioral, Psychological or Informational Intervention: Receive information about tobacco cessation
  Quality-of-Life Assessment: Ancillary studies
- VST (Virtual Counseling Sessions, NRT): Virtual Sustained Treatment (VST) patients receive an initial virtual counseling session with a study-designated tobacco treatment coach via MGH TeleHealth over 40 minutes and up to 10 more virtual counseling sessions over 15 minutes for approximately 6 months. Patients also receive up to 12 weeks of NRT (patch and lozenge combined or alone).
  Nicotine Replacement: Given NRT patch or lozenge (or both)
  Quality-of-Life Assessment: Ancillary studies
  Survey Administration: Ancillary studies
  Tobacco Cessation Counseling: Receive virtual tobacco cessation counseling
Period: Overall Study
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Started | 150 | 156
Baseline Survey | 150 | 156
3 Month Survey | 110 | 107
7-day Point Prevalence @3mo (Value or Imputed) | 147 | 154
6 Month Survey | 106 | 99
7-day Point Prevalence @6mo (Value or Imputed) | 143 | 148
Completed | 106 | 99
Not Completed | 44 | 57
Not completed — Death | 6 | 6
Not completed — Withdrawal by Subject | 7 | 18
Not completed — Lost to Follow-up | 31 | 33

BASELINE CHARACTERISTICS:
Groups:
- VST (Virtual Counseling Sessions, NRT): Virtual Sustained Treatment (VST) patients receive an initial virtual counseling session with a study-designated tobacco treatment coach via MGH TeleHealth over 40 minutes and up to 10 more virtual counseling sessions over 15 minutes for approximately 6 months. Patients also receive up to 12 weeks of NRT (patch and lozenge combined or alone).
  Nicotine Replacement: Given NRT patch or lozenge (or both) Quality-of-Life Assessment: Ancillary studies Survey Administration: Ancillary studies Tobacco Cessation Counseling: Receive virtual tobacco cessation counseling
  Survey Administration: Ancillary studies
  Tobacco Cessation Counseling: Receive virtual tobacco cessation counseling
- Total: Total of all reporting groups
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT) | Total
Number analyzed (Participants) | 150 | 156 | 306
Age, Continuous [Median (Full Range); unit: years] | 57 [27 to 81] | 57 [23 to 77] | 57 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 111 | 217
  Male | 44 | 45 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 142 | 147 | 289
  Unknown or Not Reported | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 129 | 135 | 264
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 7 | 11
Living with a smoker [Count of Participants; unit: Participants]
  Yes | 78 | 68 | 146
  No | 71 | 87 | 158
  Not reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Biochemically-confirmed 7-day Point Prevalence Abstinence at 6 Months (Not Evaluated)
Description: We will define 7-day point-prevalence by saliva cotinine (< 15 ng/ml) or expired air CO (<10 ppm). All participants who report being quit and no NRT or e-cigarette use will be requested to provide saliva samples, expired air CO will be measured in participants who report being quit and report concurrent NRT or e-cigarette use. If a participant is lost to follow-up or does not provide a saliva or CO sample, they will be considered a current smoker.
  COVID-19 restrictions prevented any saliva or CO sample collection. Therefore no biochemical outcome results are available for reporting for this aim.
Time Frame: At 6 months
Population: Due to COVID-19 restrictions saliva and CO samples could not be collected. Biochemical outcome data is not available for analysis.
Groups:
- VST (Virtual Counseling Sessions, NRT): Virtual Sustained Treatment (VST) patients receive an initial virtual counseling session with a study-designated tobacco treatment coach via MGH TeleHealth over 40 minutes and up to 10 more virtual counseling sessions over 15 minutes for approximately 6 months. Patients also receive up to 12 weeks of NRT (patch and lozenge combined or alone).
  Nicotine Replacement: Given NRT patch or lozenge (or both) Quality-of-Life Assessment: Ancillary studies Survey Administration: Ancillary studies Tobacco Cessation Counseling: Receive virtual tobacco cessation counseling
  Quality-of-Life Assessment: Ancillary studies
  Survey Administration: Ancillary studies
  Tobacco Cessation Counseling: Receive virtual tobacco cessation counseling
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Biochemically-confirmed 7-day Point Prevalence Abstinence at 3 Months (Not Evaluated)
Description: We will define 7-day point-prevalence by saliva cotinine (< 15 ng/ml) or expired air CO (<10 ppm). All participants who report being quit and no NRT or e-cigarette use will be requested to provide saliva samples, expired air CO will be measured in participants who report being quit and report concurrent NRT or e-cigarette use. If a participant is lost to follow-up or does not provide a saliva or CO sample, they will be considered a current smoker.
  COVID-19 restrictions prevented any saliva or CO sample collection or analysis as part of this study. Therefore, no biochemical outcome results are available for reporting for this aim.
Time Frame: At 3 months
Population: as for outcome 1
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: 7-day Point-prevalence Tobacco Abstinence at 6 Months - Self Report
Description: 7-day point-prevalence was determined from participant response to the survey question: "How long has it been since you last smoked a cigarette (even one or two puffs)?" If participants withdrew, was lost to follow up, did not answer, or indicated 7 days or less since their last puff, they were marked as having recently smoked.
Time Frame: At 6 months
Population: If participants withdrew, was lost to follow up, did not answer, or indicated 7 days or less since their last puff, they were marked as having recently smoked.
Measure: Count of Participants; unit: Participants
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 143 | 148
Participants | 21 | 42
Statistical Analysis 1: Comparison: EUC (Smoking Assessment, Quitting Advice, Quitline Referral) vs VST (Virtual Counseling Sessions, NRT); For self-reported 7-day point prevalence abstinence at 6-months, with a sample size of 140 in each arm then smallest detectable difference will be 22% with 80% power. Subsequent analyses will use a Bonferroni corrected alpha of 0.002 using with an estimated control rate of 31%. The primary analysis will be performed from an intent-to-treat perspective. Chi-square tests will be used to compare the outcomes between treatment groups; Test type: Equivalence — the smallest detectable difference will be 22%; p = 0.0046, Chi-squared — No correction for multiple comparisons; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.28 to 4.13]

4. Secondary Outcome: 7-day Point-prevalence Tobacco Abstinence at 3 Months - Self Report
Description: as for outcome 3
Time Frame: At 3 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 147 | 154
Participants | 22 | 38
Statistical Analysis 1: Comparison: EUC (Smoking Assessment, Quitting Advice, Quitline Referral) vs VST (Virtual Counseling Sessions, NRT); 7-day point prevalence abstinence at 3-months, with a sample size of 140 in each arm then smallest detectable difference will be 18% with 80% power and a Bonferroni corrected alpha of 0.002 using and an estimated control rate of 20%; Test type: Equivalence — the smallest detectable difference will be 22% with 80% power and a Bonferroni corrected alpha of 0.002 using and an estimated control rate of 28%; p = 0.035, Chi-squared; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.04 to 3.33]

5. Secondary Outcome: Self-reported Continuous Tobacco Abstinence
Description: Continued cessation of cigarette use was analyzed by comparing 3- and 6-month 7-day point prevalence in smoking cessation.
  If participants withdrew or did not answer the survey, they were marked as having recently smoked. Thus, participants needed to complete the survey and indicate that they had stopped tobacco use at both 3- and 6-month timepoints to be identified as having continuous cessation.
Time Frame: At 3months and 6 months
Population: If participants withdrew or did not answer the survey at the specified timepoint, they were marked as having recently smoked Analysis only includes participants having a result for the 6-month timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 143 | 148
Participants | 13 | 28
Statistical Analysis 1: Comparison: EUC (Smoking Assessment, Quitting Advice, Quitline Referral) vs VST (Virtual Counseling Sessions, NRT); power calculations assumed a sample size of 140 in each arm and a Bonferroni corrected alpha of 0.002 and an estimated control rate of 20%; Test type: Equivalence — the smallest detectable difference will be 21% with 80% power and a Bonferroni corrected alpha of 0.002 and an estimated control rate of 20%; p = 0.016, Chi-squared

6. Secondary Outcome: Sustained Tobacco Abstinence at 6 Months (Not Evaluated)
Description: To qualify as a sustained abstinence at 6 months, the participant must qualify as biochemically-verified 7-day point prevalence cigarette abstinence at 3 and 6 months. Chi-square tests will be used to compare the outcomes between treatment groups.
  COVID-19 restrictions prevented any saliva or CO sample collection. Therefore no biochemical outcome results are available for reporting for this aim.
Time Frame: At 6 months
Population: Due to COVID-19 restrictions saliva and CO samples could not be collected
Groups:
- EUC (Smoking Assessment, Quitting Advice, Quitline Referral): Patients receive an assessment of smoking status and provision of quitting advice through the screening and referral process, and are referred to the NCI Smoking Quitline.
  Behavioral, Psychological or Informational Intervention: Receive information about tobacco cessation
  Quality-of-Life Assessment: Ancillary studies
- VST (Virtual Counseling Sessions, NRT): Patients receive an initial virtual counseling session with a study-designated tobacco treatment coach via MGH TeleHealth over 40 minutes and up to 10 more virtual counseling sessions over 15 minutes for approximately 6 months. Patients also receive up to 12 weeks of NRT (patch and lozenge combined or alone).
  Nicotine Replacement: Given NRT patch or lozenge (or both)
  Quality-of-Life Assessment: Ancillary studies
  Survey Administration: Ancillary studies
  Tobacco Cessation Counseling: Receive virtual tobacco cessation counseling
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Significant Reduction in Smoking
Description: Significant reduction in daily smoking from baseline to 6 months was defined as > 50% reduction in reported number of cigarettes per day.
  Patients were ask to report the average number of cigarettes smoked per day on the 6mo and baseline surveys.
  if Xb is the average number smoked at baseline and X6 is the average number smoked at 6 months Then the reduction was calculated as (Xb-X6)/Xb
Time Frame: baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 143 | 148
Participants | 47 | 64
Statistical Analysis 1: Comparison: EUC (Smoking Assessment, Quitting Advice, Quitline Referral) vs VST (Virtual Counseling Sessions, NRT); Test type: Equivalence — no margin; p = 0.069, Chi-squared

8. Secondary Outcome: Significant Reduction in Smoking @ 3 Months
Description: Significant reduction in daily smoking from baseline to 6 months was defined as > 50% reduction in reported number of cigarettes per day.
  Patients were ask to report the average number of cigarettes smoked per day on the 3mo and baseline surveys.
  if Xb is the average number smoked at baseline and X3 is the average number smoked at 3 months Then the reduction was calculated as (Xb-X3)/Xb
Time Frame: baseline and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 147 | 154
Participants | 53 | 57
Statistical Analysis 1: Comparison: EUC (Smoking Assessment, Quitting Advice, Quitline Referral) vs VST (Virtual Counseling Sessions, NRT); Test type: Equivalence — no margin; p = 0.86, Chi-squared

9. Other Pre Specified Outcome: Potential Effect of Sociodemographics on Treatment Effectiveness
Description: Will test the effects of potential moderator in logistic regression models to determine association with tobacco abstinence. Once a parsimonious multivariate model is developed, treatment arm will be included to test for the effect of the intervention on the moderator. Interactions between the treatment arm and the moderators to indicate the relationship between the moderators and the treatment group on the effectiveness outcomes. Also, generalized estimating equations (GEE) will be used to look at longitudinal models. Multiple comparisons will be accounted for by considering Bonferroni adjustments.
Time Frame: Up to 6 months
Reporting Status: Not Posted, anticipated posting 2025-06

10. Other Pre Specified Outcome: Potential Effect of Medical and Smoking History on Treatment Effectiveness
Description: as for outcome 9
Time Frame: Up to 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Potential Effect of Cancer Variables on Treatment Effectiveness
Description: as for outcome 9
Time Frame: Up to 6 months
Reporting Status: Not Posted, anticipated posting 2025-06

12. Other Pre Specified Outcome: Implementation of the Intervention at Community Oncology Sites
Description: Will follow Proctor and colleagues' recommended taxonomy for measurement of implementation outcomes. Will measure acceptability (satisfaction with content/delivery), adoption (program uptake), appropriateness (relevance), cost, and treatment fidelity/adaptation and penetration (reach) and sustainability. These implementation outcomes will be assessed with mixed methods using qualitative and quantitative data to be collected from patient, tobacco treatment counselor, NCORP oncology principal investigators (PIs) and provider clinicians/staff, and electronic health record (EHR) documentation. Will use descriptive statistics to summarize implementation outcomes (acceptability, adoption, appropriateness, fidelity, cost, penetration and sustainability) and conduct treatment group comparisons (i.e., acceptability).
Time Frame: Up to 36 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Intervention Acceptability (Satisfaction With Content/Delivery) at Community Oncology Sites
Description: Outcome will be assessed with mixed methods using qualitative & quantitative data to be collected from patient, tobacco treatment counselor, NCORP oncology principal investigators (PIs) and provider clinicians/staff, and electronic health record (EHR) documentation. Will use descriptive statistics to summarize implementation outcome and conduct treatment group comparisons.
Time Frame: Up to 36 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Intervention Adoption (Program Uptake) at Community Oncology Sites
Description: as for outcome 13
Time Frame: Up to 36 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Intervention Appropriateness (Relevance) at Community Oncology Sites
Description: as for outcome 13
Time Frame: Up to 36 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Intervention Cost at Community Oncology Sites
Description: as for outcome 13
Time Frame: Up to 36 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Treatment Fidelity/Adaptation at Community Oncology Sites
Description: as for outcome 13
Time Frame: Up to 36 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Intervention Penetration (Reach) at Community Oncology Sites
Description: as for outcome 13
Time Frame: Up to 36 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Intervention Sustainability at Community Oncology Sites
Description: as for outcome 13
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2025-06

20. Other Pre Specified Outcome: Acceptability: Needs Were Met
Description: Guided by Proctor and colleagues' (2011) recommendations for measurement of implementation outcomes, we will explore Patient satisfaction with content/delivery of their randomly assigned tobacco treatment (acceptability) to gain an initial understanding of the implementation process.
  Results of the responses to the "To what extent has the Smoke Free Support Study program met your needs?" acceptability question on the 6-month questionnaire rating from 1 (None of my needs have been met) to 4 (Almost all of my needs have been met) with higher scores indicating more needs met.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Groups:
- Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral): Patients receive an assessment of smoking status and provision of quitting advice through the screening and referral process, and are referred to the NCI Smoking Quitline.
  Behavioral, Psychological or Informational Intervention: Receive information about tobacco cessation
  Quality-of-Life Assessment: Ancillary studies
- Virtual Counseling (Virtual Counseling Sessions, NRT): Patients receive an initial virtual counseling session with a study-designated tobacco treatment coach via MGH TeleHealth over 40 minutes and up to 10 more virtual counseling sessions over 15 minutes for approximately 6 months. Patients also receive up to 12 weeks of NRT (patch and lozenge combined or alone).
  Nicotine Replacement: Given NRT patch or lozenge (or both)
  Quality-of-Life Assessment: Ancillary studies
  Survey Administration: Ancillary studies
  Tobacco Cessation Counseling: Receive virtual tobacco cessation counseling
Arm/Group | Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral) | Virtual Counseling (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 99 | 89
Participants
  None of my needs have been met | 25 | 4
  Only a few of my needs have been met | 37 | 9
  Most of my needs have been met | 24 | 38
  Almost all of my needs have been met | 12 | 37
  Skipped question | 1 | 1
Statistical Analysis 1: Comparison: Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral) vs Virtual Counseling (Virtual Counseling Sessions, NRT); Fisher's exact tests were performed to assess the differences between the VST and EUC arms on the 6-month questionnaire; Test type: Equivalence — No equivalence margin; p < .0001, Fisher Exact — Alpha level 0.01

21. Other Pre Specified Outcome: Acceptability: Assistance Support
Description: Guided by Proctor and colleagues' (2011) recommendations for measurement of implementation outcomes, we will explore Patient satisfaction with content/delivery of their randomly assigned tobacco treatment (acceptability) to gain an initial understanding of the implementation process.
  Results of the responses to the "Did you get the kind of smoking cessation assistance that you wanted?" acceptability question on the 6-month questionnaire rating from 1 (No, definitely not) to 4 (Yes, definitely) with higher scores indicating greater confidence that assistance met desired level.
Time Frame: 6-months
Population: Only patients answering the acceptability question are reported
Measure: Count of Participants; unit: Participants
Groups:
- EUC (Smoking Assessment, Quitting Advice, Quitline Referral): Enhanced Usual Care patients receive an assessment of smoking status and provision of quitting advice through the screening and referral process, and are referred to the NCI Smoking Quitline.
  Behavioral, Psychological or Informational Intervention: Receive information about tobacco cessation
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | EUC (Smoking Assessment, Quitting Advice, Quitline Referral) | VST (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 99 | 89
Participants
  No, definitely not | 16 | 2
  No, not really | 43 | 7
  Yes, generally | 35 | 40
  Yes, definitely | 5 | 40
Statistical Analysis 1: Comparison: EUC (Smoking Assessment, Quitting Advice, Quitline Referral) vs VST (Virtual Counseling Sessions, NRT); Fisher's exact tests were performed to assess the differences between the VST and EUC arms on the 6-month questionnaire; Test type: Equivalence — No equivalence margin; p < .0001, Fisher Exact — Alpha level 0.01

22. Other Pre Specified Outcome: Acceptability: Helpfulness of Study
Description: Guided by Proctor and colleagues' (2011) recommendations for measurement of implementation outcomes, we will explore Patient satisfaction with content/delivery of their randomly assigned tobacco treatment (acceptability) to gain an initial understanding of the implementation process.
  Results of the responses to the "How helpful has the Smoke Free Support Study been for you?" acceptability question on the 6-month questionnaire rating from 1 (Not at all helpful) to 5 (Very helpful) with higher scores indicating increased helpfulness.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral) | Virtual Counseling (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 99 | 89
Participants
  Not at all helpful | 17 | 3
  Not very helpful | 17 | 1
  Neutral | 31 | 10
  Somewhat helpful | 23 | 31
  Very helpful | 11 | 44
Statistical Analysis 1: Comparison: Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral) vs Virtual Counseling (Virtual Counseling Sessions, NRT); Fisher's exact tests were performed to assess the differences between the VST and EUC arms on the 6-month questionnaire; Test type: Equivalence — No equivalence margin; p < .0001, Fisher Exact — Alpha level 0.01

23. Other Pre Specified Outcome: Acceptability: Quality of Assistance
Description: Guided by Proctor and colleagues' (2011) recommendations for measurement of implementation outcomes, we will explore Patient satisfaction with content/delivery of their randomly assigned tobacco treatment (acceptability) to gain an initial understanding of the implementation process.
  Results of the responses to the "How would you rate the quality of the smoking cessation assistance that you received?" acceptability question on the 6-month questionnaire rating from 1 (Poor) to 4 (Excellent) with higher scores indicating more greater quality
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral) | Virtual Counseling (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 99 | 89
Participants
  Did not answer | 1 | 1
  Poor | 20 | 2
  Fair | 38 | 3
  Good | 30 | 39
  Excellent | 10 | 44

24. Other Pre Specified Outcome: Acceptability: Would Recommend Study to Friends
Description: Guided by Proctor and colleagues' (2011) recommendations for measurement of implementation outcomes, we will explore Patient satisfaction with content/delivery of their randomly assigned tobacco treatment (acceptability) to gain an initial understanding of the implementation process.
  Results of the responses to the "If a friend were in need of similar help, would you recommend the Smoke Free Support Study to him or her?" acceptability question on the 6-month questionnaire Ratings from 1 (No, definitely not) to 4 (Yes, definitely) with higher scores indicating more greater likelihood of recommending.
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral) | Virtual Counseling (Virtual Counseling Sessions, NRT)
Number analyzed (Participants) | 99 | 89
Participants
  No, definitely not | 3 | 1
  No, I don't think so | 23 | 4
  Yes, I think so | 50 | 32
  Yes, definitely | 19 | 51
  Did Not Answer | 4 | 1
Statistical Analysis 1: Comparison: Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral) vs Virtual Counseling (Virtual Counseling Sessions, NRT); Fisher's exact tests were performed to assess the differences between the VST and EUC arms on the 6-month questionnaire; Test type: Equivalence — No equivalence margin; p < .0001, Fisher Exact — Alpha level 0.01

ADVERSE EVENTS:
Time Frame: from randomization up to 1 year
Description: Adverse events were only reportable for subjects on the Virtual Intervention arm of the study (ie., those with the possibility of being recommended Nicotine Replacement Therapy from the study team)
Arm/Group | Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral) | Virtual Counseling (Virtual Counseling Sessions, NRT)
All-Cause Mortality (participants affected / at risk) | 13/150 | 10/156
Serious Adverse Events (participants affected / at risk) | 13/150 | 10/156
Other Adverse Events (participants affected / at risk) | 0/150 | 0/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Usual Care (Smoking Assessment, Quitting Advice, Quitline Referral) (N=150) | Virtual Counseling (Virtual Counseling Sessions, NRT) (N=156)
Death, NOS (General disorders) | 6 (6) | 4 (4)
Other (General disorders) | 5 (5) | 2 (2) — Other Unspecified
Disease progression (Renal and urinary disorders) | 2 (2) | 2 (2) — Death, Renal Cell Carcinoma disease progression
Cardiac Arrest (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03808818/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03808818/ICF_001.pdf